CLINICAL TRIAL: NCT03426865
Title: Anti-1-amino-3-18F-flurocyclobutane-1-carboxylic Acid (Axumin) Positron Emission Tomography/Computed Tomography Prior to Retroperitoneal Lymph Node Dissection for Testicular Cancer
Brief Title: Role of Axumin PET Scan in Germ Cell Tumor
Acronym: TESTPET
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, yair lotan, Professor of Urology, University of Texas Southwestern Medical Center
Other Study IDs: STU 032017-051
Record Dates: First submitted 2018-01-25; First posted 2018-02-08 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Testis Cancer; Germ Cell Tumor; Testicular Cancer; Germ Cell Tumor of Testis; Germ Cell Tumor, Testicular, Childhood; Testicular Neoplasms; Testicular Germ Cell Tumor; Testicular Yolk Sac Tumor; Testicular Choriocarcinoma; Testicular Diseases; Germ Cell Cancer Metastatic; Germ Cell Neoplasm of Retroperitoneum; Germ Cell Cancer, Nos
Keywords: retroperitoneal lymph node dissection; testicular cancer; testis cancer; germ cell tumor; PET scan; Axumin; teratoma
MeSH Terms: conditions — Testicular Neoplasms; Neoplasms, Germ Cell and Embryonal; Testicular Germ Cell Tumor; Endodermal Sinus Tumor; Testicular Diseases; Teratoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Axumin PET scan: Only one arm is being evaluated--the arm receiving PET scan
  Interventions: Drug: Axumin PET scan

INTERVENTIONS:
Drug: Axumin PET scan — PET scan prior to RPLND
  Other Names: PET SCAN ARM

SUMMARY:
Investigators will use Axumin PET/CT to help with the imaging modalities to determine the presence of occult retroperitoneal disease.

DETAILED DESCRIPTION:
Investigators aim to perform a prospective study of anti-18F-FACBC PET/CT in patients with NSGCT prior to RPLND, either in the primary setting or in the post-chemotherapy setting. We will correlate histopathologic outcomes from the RPLND specimen and clinical outcomes of recurrence during follow-up to identify the accuracy of anti-18F-FACBC PET/CT in these settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed NSGCT after orchiectomy who are scheduled to undergo primary RPLND or post-chemotherapy RPLND
* Patients must be over 18 years old and capable and willing to provide informed consent.
* Medically stable as judged by patient's physician.
* Life expectancy must be estimated at > 6 months.
* Patients must have an ECOG performance status of 0-3 (restricted to ECOG PS 0-2 if age >70 years).
* Patient must be able to lie still for a 20 to 30 minute PET/CT scan. Patients will be asked if they have problems or issues with lying flat

Exclusion Criteria:

* Patients with known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals of similar chemical or biologic composition to anti-18F-FACBC are NOT eligible.
* Patients with liver failure are NOT eligible.
* Patients currently undergoing chemotherapy or chemotherapy within two weeks of anti-18F-FACBC PET/CT scan are NOT eligible

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males with germ cell tumors (testicular cancer)
Study Population: Population will be selected from patients seen in the clinic at University of Texas Southwestern Medical Center
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Performance characteristics of Axumin PET scan in patients undergoing retroperitoneal lymph node dissection | Two years
  Investigate the accuracy of anti-18F-FACBC PET/CT correlating with histopathologic outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Yair Lotan, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No